CLINICAL TRIAL: NCT05029570
Title: Conduction System PACing and Atrioventricular Node Ablation in Patients With hEart Failure, Left Ventricular Ejection Fraction >40% and Permanent Atrial FIBrilation: the PACE-FIB Trial
Brief Title: Heart Rate Regularization in Atrial Fibrilation and Heart Failure
Acronym: PACE-FIB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Rodríguez Muñoz (Other)
Collaborators: Sociedad Castellana de Cardiologia (Other)
Responsible Party: Sponsor-Investigator, Daniel Rodríguez Muñoz, Consultant in Cardiac Electrophysiology, Principal Investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PACE-FIB
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: atrial fibrillation;; heart failure;; conduction system pacing;; heart rate regularization
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Medical Device: Conduction System Pacing (pacemaker implantation)
Who Masked: Outcomes Assessor
Masking Description: Clinical outcomes will be adjudicated by the investigator and reviewed by the Clinical Events Committee, that will be blind to treatment received by the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conduction System Pacing and AV node ablation (Experimental): Atrioventricular node ablation and subsequent conduction system pacing
  Interventions: Device: Conduction System Pacing (pacemaker implantation)
- Medical treatment for rate control of AF (No Intervention): Pharmacological rate control based on clinical practice guidelines

INTERVENTIONS:
Device: Conduction System Pacing (pacemaker implantation) — Conduction System Pacing (pacemaker implantation) and Atrioventricular node ablation
  Other Names: Atrioventricular node ablation
  Arms: Conduction System Pacing and AV node ablation

SUMMARY:
The PACE-FIB trial is a multicentre, randomised, open-label clinical trial. Patients older than 18 years, with permanent AF, LVEF>40%, average resting heart rate ≤ 110 beats per minute (bpm), at least one hospitalisation due to HF in the previous year and basal NT-proBNP level>900 pg/ml will be randomised to either CSP and subsequent AV node ablation (intervention group) vs. pharmacologic rate control optimised according to clinical practice guidelines. The impact of both strategies on a composite primary endpoint of all-cause mortality, HF hospitalisation and worsening HF will be evaluated during a 36-month follow-up.

DETAILED DESCRIPTION:
Permanent atrial fibrillation (AF) causes beat-to-beat heart rate irregularity, which has shown to decrease cardiac output. Observational data suggest that heart rate regularization through atrioventricular (AV) node ablation and pacemaker implantation improves outcomes in heart failure (HF) patients. However, no trials have been conducted to assess its potential benefit in HF and left ventricular ejection fraction (LVEF)>40%, a population in whom treatment strategies effectively improving outcomes are scarce.

The goal of this trial is to assess the benefit of heart rate regularization through AV node ablation and conduction system pacing (CSP) in patients with permanent AF and HF with preserved or mildly reduced systolic function. The investigators hypothesize that heart rate regularization added to physiological pacing - preventing the deleterious effect of right apical pacing - reduces mortality, HF hospitalisations or worsening HF in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Permanent atrial fibrillation
* At least one episode of hospitalisation due to heart failure in the previous 12 months.
* Left ventricular ejection fraction > 40%
* Average resting heart rate ≤ 110 beats per minute
* NT-proBNP ≥ 900 pg/ml in the 30 days prior to enrollment
* Age ≥ 18 years
* Capacity to understand the nature of the study, legal ability and willingness to give informed consent.

Exclusion Criteria:

* Severe frailty (Clinical Frailty Scale ≥ 7) or comorbidity reducing life expectancy to < 12 months.
* Acute heart failure at the time of enrollment or systolic blood pressure < 80 mmHg in the absence of inotropic agents.
* Severe chronic kidney disease (estimated Glomerular Filtration Rate ≤ 20 ml/1,73 m2
* Severe mitral or aortic valvular heart disease
* Anaemia (Haemoglobin < 10 g/dl)
* Morbid obesity (BMI ≥ 35)
* Severe Chronic Obstructive Pulmonary Disease (Gold ≥ 3)
* Presence of a different indication for pacing of implantable cardioverter-defibrillator (ICD)
* Obstructive hypertrophic cardiomyopathy
* Infiltrative cardiomyopathy (amyloidosis, sarcoidosis, Fabry disease, others)
* Simultaneous participation in a different trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint | 36 months
  All-cause mortality, heart failure hospitalisation and worsening heart failure

SECONDARY OUTCOMES:
All-cause mortality | 36 months
  Mortality due to any cause
Cardiovascular mortality | 36 months
  Mortality due to cardiovascular causes
Heart failure hospitalization | 36 months
  Hospitalization due to heart failure decompensation
Worsening heart failure | 36 months
  An episode of heart failure diagnosed based on symptoms, signs, imaging and analytical criteria that requires unplanned medical attention and intravenous diuretic therapy
Unplanned cardiovascular hospitalisation | 36 months
  Unplanned cardiovascular hospitalisation
Left ventricular ejection fraction | 12 months
  assessed by the Simpson method
Change in left ventricular dimension | 12 months
  end-diastolic and end-systolic volumes
Change in degree of mitral regurgitation | 12 months
  Change in degree of mitral regurgitation
Change in functional status | 36 months
  Assessed by New York Heart Association (NYHA) on a I to IV scale (I being better functional status and IV worst possible functional status)
Major adverse events during or in the first 30-days following pacemaker implantation | 30 days
  Percentage of patients suffering one of the following: death, cardiac tamponade, perforation requiring cardiac surgery, pneumothorax, haemothorax, device infection, endocarditis, lead displacement requiring re-intervention
Major adverse events during or in the first 30-days following atrioventricular node ablation | 30 days
  Percentage of patients suffering one of the following: death, cardiac tamponade, perforation requiring cardiac surgery, puncture site vascular complications requiring vascular surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Arribas Ynsaurriaga, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No